CLINICAL TRIAL: NCT06365177
Title: Evaluation of the Concordance of Five Times Sit To Stand Results Between a Physical Consultation and a Teleconsultation of the Elderly
Brief Title: Evaluation of the Concordance of Five Times Sit To Stand Results Between a Physical Consultation and a Teleconsultation
Acronym: TELETEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 29BRC22.0243
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Rehabilitation; Elderly Person; Teleconsultation
Keywords: Five Time Sit To Stand; Teleconsultation
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Intervention Model Description: Cross-sectional interventional multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical consultation followed by Teleconsultation (Other): First, patients take the Five Time Sit To Stand in the presence of the physiotherapist. Then, patients perform the test in a room away from the physiotherapist (there are a computer with a webcam is set up on a desk).
  There will be a 5-minute rest period between the 2 test conditions (physical consultation and teleconsultation).
  Each test is performed 2 times. The best time will be retained for analysis.
  Interventions: Other: Physical consultation; Other: Teleconsultation
- Teleconsultation followed by physical consultation (Other): First, patients perform the Five Time Sit To Stand in a room away from the physiotherapist (there are a computer with a webcam is set up on a desk). Then, patients take the test in the presence of the physiotherapist. There will be a 5-minute rest period between the 2 test conditions (teleconsultation and physical consultation).
  Each test is performed 2 times. The best time will be retained for analysis.
  Interventions: Other: Physical consultation; Other: Teleconsultation

INTERVENTIONS:
Other: Physical consultation — The subject enters a room where the therapist is present. A chair is placed against a wall in the same room.
  Once again, the therapist suggests repeating the test. During the test, the therapist sits opposite the patient, at the same distance as the computer used during the teleconsultation.
Other: Teleconsultation — Prior to the test, the investigator should carry out a "mock" test with a volunteer from the facility, for example, to ensure wifi, sound and image functionality.
  The patient enters a room where a computer equipped with a webcam is set up on a desk. The teleconsultation has already started when the patient enters the room. No recordings are made.
  A chair is placed at a distance from the desk, with the backrest against a wall. The chair faces the computer. The desk or table where the computer is located is about 3 meters from the participant, ensuring that the webcam can frame the patient's entire body during the test.
  With the consultation already underway, the investigator can direct the patient to sit in the chair against the wall. The investigator will make sure that the patient hears the instructions given.
  Once the patient is seated on the chair, the therapist explains the test procedure and shows it once to make sure the subject understands it.

SUMMARY:
This study concerns elderly person aged more than 65 years with autonomous mobility.

It is a multicentric randomized trial in two arms :

Arm one : remote consultation then physical consultation Arm two : physical consultation then remote consultation

Consultations consist to take a Five Times Sit To Stand test, in physical consultation with physiotherapist in the same room and in remote consultation with a physiotherapist in the next room to the patient.

DETAILED DESCRIPTION:
This study concerns elderly person aged more than 65 years with autonomous mobility.

It is a multicentric randomized trial in two arms :

Arm one : remote consultation then physical consultation Arm two : physical consultation then remote consultation

Consultations consist to take a Five Times Sit To Stand test, in physical consultation with physiotherapist in the same room and in remote consultation with a physiotherapist in the next room to the patient.

Tests are realized at baseline after randomization. The test with best time will be considered for analysis.

Once the 2 tests have been carried out, a satisfaction survey will evaluate the preference between the two tests for each patient.

Patients will be re-contacted by telephone at 3, 6 and 12 months post-inclusion to collect the number of falls.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over the age of 65.
* Elderly people who can walk and move around independently.
* Subjects capable of giving informed consent.
* GIR 3,4,5,6.
* Affiliated to a Social Security scheme.

Exclusion Criteria:

* GIR < 3
* Major visual and/or hearing impairment (known pathology and not fitted with hearing aids)
* Patient deprived of liberty by judicial or administrative decision, under guardianship or curatorship
* Subject having refused to participate.
* Subject at risk of syncope on rising (cardiac pathologies, orthostatic hypotension).
* Subjects with known vestibular disorders.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Five Time Sit To Stand test completion time in teleconsultation | At inclusion
  The physiotherapist is present in a room at a distance from the patient's consultation room.
  The Five Time Sit to Stand (FTSS) is a functional assessment that requires a chair and a stopwatch. The patient is timed from start to finish. The time taken to complete the test is expressed in minutes.
  The patient performs two trials. The best result is retained for analysis.
Five Time Sit To Stand test completion time in face-to-face consultation | At inclusion
  The physiotherapist is present in the same consulting room as the patient. The Five Time Sit to Stand (FTSS) is a functional assessment that requires a chair and a stopwatch. The patient is timed from start to finish. The time taken to complete the test is expressed in minutes.
  The patient performs two trials. The best result is retained for analysis.

SECONDARY OUTCOMES:
Satisfaction questionnaire | At inclusion
  It is a questionnaire with 4 questions:
  Question n°1 : 3 answers Question n°2 : bimodal response (Yes /No) Question n°3 : 5 answers Question n°4 : 4 answers
  Moreover, the therapist completes the following question for each patient:
  - Do you think this patient could benefit from a follow-up by performing the same test in teleconsultation at home? Yes/No
Five Time Sit To Stand test completion time in teleconsultation | At inclusion
  The physiotherapist is present in a room at a distance from the patient's consultation room.
  The Five Time Sit to Stand (FTSS) is a functional assessment that requires a chair and a stopwatch. The patient is timed from start to finish. The time taken to complete the test is expressed in minutes.
  The patient performs two trials. The best result is retained for analysis.
Five Time Sit To Stand test completion time in face-to-face consultation | At inclusion
  The physiotherapist is present in the same consulting room as the patient. The Five Time Sit to Stand (FTSS) is a functional assessment that requires a chair and a stopwatch. The patient is timed from start to finish. The time taken to complete the test is expressed in minutes.
  The patient performs two trials. The best result is retained for analysis.
Presence or absence of falls | At Month 3, Month 6 and Month 12
  Phone call to ask if patient has fallen (Yes/No)
Number of falls | At Month 3, Month 6 and Month 12
  Phone calls to ask the number of falls.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - ILDYS Ty Yann, Brest
  - Institut de réadaptation du Cap Horn, Landerneau

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.